CLINICAL TRIAL: NCT03955276
Title: An Open Label Navigational Investigation of Molecular Profile-Related Evidence Determining Individualized Cancer Therapy for Patients With Incurable Hematologic Malignancies and Poor Prognoses (I-PREDICT Heme)
Brief Title: An Open Label Navigational Investigation of Molecular Profile-Related Evidence Determining Individualized Cancer Therapy for Patients With Incurable Hematologic Malignancies (I-PREDICT Heme)
Acronym: I-PREDICT Heme
Status: Terminated | Type: Observational
Why Stopped: PI left the institution.
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: 181350
Record Dates: First submitted 2019-04-01; First posted 2019-05-20 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Hematologic Cancer
Keywords: Hodgkin lymphoma; non-Hodgkin lymphoma; Acute leukemia; Chronic leukemia; rare hematologic tumors; Hematopoietic lymphoid/myeloid cancer
MeSH Terms: conditions — Hematologic Neoplasms; Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A sample of the subject's blood and/or tumor specimen will be collected during screening and prior to study treatment. The sample will be reviewed by hematopathology. Genomic /immunophenotypic studies will be performed to guide therapy selection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Matched Therapy: Targeted therapy matched to each patient's genomic/immunophenotypic tumor profile (whereby oncogenic alterations are matched with targeted agents)
  Interventions: Other: Molecularly targeted treatment matched to genomic/immunophenotypic tumor profile (chosen by treating physician)
- Unmatched Therapy: General, unmatched therapy (standard of care)

INTERVENTIONS:
Other: Molecularly targeted treatment matched to genomic/immunophenotypic tumor profile (chosen by treating physician) — Biologically targeted matched treatment (chosen by treating physician)
  Groups: Matched Therapy

SUMMARY:
The purpose of this study is to perform a prospective study that is histology-independent personalized navigation approach to cancer therapy based upon tumor molecular profile as determined by Clinical Laboratory Improvement Amendments (CLIA) certified comprehensive genomic analysis. The molecular mutation profile will then be matched to existing, FDA-approved, targeted agents or to existing clinical trials using investigational agents for treatment of patients with incurable hematologic malignancies for whom no effective standard therapy exists or who have either exhausted or are intolerant of standard options.

ELIGIBILITY:
Inclusion Criteria:

* Patients with incurable hematologic malignancies with ≥50% 2-year cancer-associated mortality.
* Patients with relapsed/refractory hematologic malignancies, irrespective of 2-year mortality, who, in the opinion of the investigator, have no treatment option expected to yield significant clinical benefit.
* Patients with a rare tumor histology (i.e., fewer than 6 cases per 100,000 per year) with no approved therapies.
* Patients must have measurable disease for malignancies: defined as at least one lesion that can be accurately measured in at least one dimension with spiral CT scan, PET-CT, MRI, or calipers by clinical exam. Or presence of hematologic abnormalities with or without bone marrow involvement.
* Patients must have evaluable tissue/blood with adequate tumor content/purity for testing as specified by the molecular profiling lab. This will be obtained during the standard of care tumor diagnosis and tumor staging evaluation.
* Age ≥ 18 years.
* ECOG Performance Status 0-2.
* New York Heart Association (NYHA) Functional Classification I-II.
* Adequate organ function that reasonably allows for safe administration of therapy.
* At the time of treatment, patients should be off other anti-tumor agents for at least 5 half-lives of the agent or 2 weeks from the last day of treatment, whichever is shorter, so long as there is recovery from clinically significant side effects from previous therapy to less than or equal Grade 1.
* Able to swallow and/or retain oral medication, if needed.
* Ability to understand and the willingness to sign a written informed consent.
* Female patients of childbearing potential must agree to use at least one form of contraception during the study.

Patients must have at least one of the following for a diagnosis/disease status:

1. Advanced symptomatic disease
2. Medically unfit for standard therapy
3. Disease where no conventional therapy leads to a survival benefit > 3 months in the respective cohort and line of therapy for which the patient is otherwise eligible
4. Actionable biologically informed targets determined by certified genomic profiling, immunophenotyping or other clinically validated techniques.

Exclusion Criteria:

* Severe or uncontrolled medical disorder that would, in the investigator's opinion, confound study analyses of treatment response or preclude the patient from safely receiving treatment (i.e. substance abuse or psychiatric illness/social situations that would limit compliance with study requirements).
* Pregnancy, breast-feeding women or any patient with childbearing potential not using adequate pregnancy prevention.
* Inadequate end organ function that would preclude safe administration of anti-neoplastic therapy; including hepatic dysfunction (LFTs > 5 x normal limit, total bilirubin > 3 and Cr > 3 x normal limit or GFR < 20 cc/min, or symptomatic heart failure (EF < 20%), except when organ function impairment is a consequence of underlying malignancy and there is a reasonable expectation for improvement following initiation of appropriate therapy.
* Uncontrolled infections or sepsis. Patients with chronic viral infections (including HIV, HBV/HCV) that are controlled with appropriate concurrent therapy are allowed to participate in the study, provided ongoing compliance with antiviral therapy can be reasonably expected throughout the duration of the study. Patients with acute infections must start appropriate anti-microbial therapy and demonstrate stabilization of infection prior to study initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with incurable or relapsed/refractory hematologic malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Response rate | 3.5 years
  Assess overall response rates to molecularly targeted matched treatment and physician's choice of unmatched standard-of-care treatment.

SECONDARY OUTCOMES:
Incidence of grade 3-5 adverse event | 3.5 years
  Incidence of grade 3-5 adverse events in all groups according to CTCAE v4.03
Overall response rate (ORR) | 3.5 years
  Overall response rate (ORR) defined as partial response (PR) or complete response (CR) according to disease specific NCCN response criteria
Progression free survival (PFS) | 3.5 years
  Progression free survival (PFS) defined as time from first dose to disease progression or death whichever occurs first
Overall survival (OS) | 3.5 years
  Overall survival (OS) defined as time from first dose to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Galanina, MD, Principal Investigator — UCSD/MCC
Locations (1):
- UCSD Moore's Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No